CLINICAL TRIAL: NCT01592201
Title: An Open-label, Prospective, Randomized and Comparative Study of Patient Satisfaction Between Continued Administration of Previous Antipsychotics Versus Switched Administration to Paliperidone ER in Non-satisfied Patients With Previous Antipsychotic Drug
Brief Title: A Comparative Study of Patient Satisfaction Between Continued Administration of Previous Antipsychotics Versus Switched Administration to Paliperidone ER in Non-satisfied Patients With Previous Antipsychotic Drug
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: This study was early terminated due to insufficient enrollment required for hypothesis testing.
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR100782; PAL-KOR-4019 (Other: Janssen Korea, Ltd., Korea); R076477SCH4064 (Other: Janssen Korea, Ltd., Korea)
Record Dates: First submitted 2012-02-10; First posted 2012-05-07 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Paliperidone ER; Antipsychotics; Mental disorder; Comparative study
MeSH Terms: conditions — Schizophrenia; Mental Disorders | interventions — Aripiprazole; Olanzapine; Risperidone; Antipsychotic Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paliperidone ER (Experimental): Immediate initiation of Paliperidone ER for a total of 12 weeks
  Interventions: Drug: Paliperdidone ER
- Antipsychotics and paliperidone ER (Experimental): Delayed initiation included previous atypical antipsychotics for 8 weeks and then be initiated on paliperidone ER at Day 56 for 4 weeks. The atypical antipsychotics includes aripiprazole, olanzapine and risperidone. These antipsychotics belongs to the class of second generation bipolar atypical antipsychotics.
  Interventions: Drug: Paliperdidone ER; Drug: Aripiprazole, olanzapine and risperidone (Antipsychotics)

INTERVENTIONS:
Drug: Paliperdidone ER — Form = osmotic release oral system, route = oral
Drug: Aripiprazole, olanzapine and risperidone (Antipsychotics) — Form = tablet, route = oral
  Arms: Antipsychotics and paliperidone ER

SUMMARY:
The purpose of this study is to compare the patient satisfaction between continued administration of previous antipsychotics versus switched administration to paliperidone ER in non-satisfied patients with previous (paliperidone)

DETAILED DESCRIPTION:
This is a randomized (patients are assigned to intervention by chance), prospective, open-label (all people involved know the identity of the assigned drug), switch study designed to evaluate patient-assessed medication satisfaction after 12 weeks of treatment in patients with schizophrenia. The total duration of this study is 12 weeks. Outpatients who treated atypical antipsychotics and report dissatisfaction (Medication Satisfaction Questionnaire [MSQ] <4) with their current treatment response are eligible to participate in the study. Patients will be randomized into two groups, 1) Patients randomized to an immediate initiation of paliperidone ER for a total 12 weeks 2) Patients randomized to a delayed initiation will continue their previous atypical antipsychotics for 8 weeks and then be initiated on paliperidone ER at Day 56 for 4 weeks. During the study treatment optimization will be done by dose adjustment (dose increase or decrease) and by adding psychotropic agents except the antipsychotics.

ELIGIBILITY:
Inclusion Criteria:

* Must be diagnosed with schizophrenia according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) criteria
* Have taken atypical antipsychotics (aripiprazole, olanzapine, risperidone) at least 6 weeks prior to start of study.
* Have Medication Satisfaction Questionnaire (MSQ) score of ≤3
* Competent patients who manage to answer the questionnaires

Exclusion Criteria:

* Have had a history or current symptoms of tardive dyskinesia or neuroleptic malignant syndrome
* Have had relevant history of or current presence of any significant or unstable cardiovascular, respiratory, neurological (including seizures or significant cerebrovascular), renal, hepatic, hematologic, endocrine, immunologic, morbid obesity (BMI≥40), or other systemic disease
* Had received two or more different kind of antipsychotics.
* Had a history of taking paliperidone extended release (ER).
* Allergy or hypersensitivity to risperidone or paliperidone ER.
* Have been on clozapine or long-acting injectable antipsychotic medication during the last 3 months.
* Have had Medication Satisfaction Questionnaire (MSQ) score>3
* Have been hospitalized for longer than 8 continuous weeks during the past 6 months
* Had history of any severe preexisting gastrointestinal narrowing (pathologic or iatrogenic) or inability to swallow the oral tolerability medication whole with the aid of water for patients requiring oral tolerability testing
* Current substance dependence (DSM-IV) or past history of dependence (more than 6 months)

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-07; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in the medication satisfaction questionnaire (MSQ) score at Week 8 | Baseline and Week 8
  A single-item, global, patient-completed instrument that is read aloud to patients by clinicians designed to assess treatment satisfaction among patients with schizophrenia. It consists of one question: "Overall, how satisfied are you with your current antipsychotic medication(s)?" with responses assessed on a 7-point scale rated as follows: 1 = extremely dissatisfied, 2=very dissatisfied, 3=somewhat dissatisfied, 4=neither satisfied nor dissatisfied, 5=somewhat satisfied, 6 = very satisfied, 7 = extremely satisfied

SECONDARY OUTCOMES:
Positive and negative symptoms scale (PANSS) score | Baseline to Week 12
  The PANSS provides a total score (sum of the scores of all 30 items) and scores for 3 subscales, the positive subscale (7 items), the negative subscale (7 items), and the general psychopathology subscale (16 items), each rated on a scale of 1 (absent) to 7 (extreme). It's designed to capture symptoms of schizophrenia. (Gold standard)
Drug Attitude Inventory (DAI)-10 Score | Baseline to Week 12
  DAI-10 is a 10-item scale developed to assess how the attitude of schizophrenia patients toward their medications may affect compliance (-10~+10)
Clinical Global Impression-Severity (CGI-S) Score | Baseline to Week 12
  The CGI-S rating scale is used to rate the severity of a patient's psychotic condition on a 7-point scale ranging from 1 (not ill) to 7 (extremely severe)
Personal and Social Performance Scale (PSP) | Baseline to Week 12
  This scale assesses the degree of dysfunction a patient exhibits within 4 domains of behavior: socially useful activities, personal and social relationships, self-care, and disturbing and aggressive behavior. The score ranges from 1 to 100, divided into 10 equal intervals to rate the degree of difficulty (i, absent to vi, very severe) in each of the 4 domains. Based on the four domains there will be one total score. Patient's with a score of 71 to 100 have a mild degree of difficulty; from 31 to 70, varying degrees of disability; ≤ 30, functioning so poorly as to require intensive supervision
Sleep Visual Analog Scale (Sleep VAS) | Baseline to Week 12
  This self-administered scale rates quality of sleep and daytime drowsiness. Patient's will indicate on an 11- point scale (from 0 to 10) how well they have slept in the previous 7 days ("very badly" to "very well") and how often they have felt drowsy within the previous 7 days ("not at all" to "all the time"). On the sleep evaluation scale, score '0' corresponds to 'very badly' and score '10' to 'very well'. On the daytime drowsiness scale, score '0' corresponds to 'not at all' and score '10' to 'all the time
Number of patients with adverse events | Baseline to Week 12
Number of patients with vital signs and physical examination | Baseline to Week 12
Number of patients with laboratory test (prolactin, blood glucose, glycosylated hemoglobin, cholesterol, triglyceride) | Baseline to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd., Korea Clinical Trial, Study Director — Janssen Korea, Ltd., Korea
Locations (9):
- South Korea (9):
  - Busan
  - Cheonan
  - Chuncheon
  - Chungju
  - Daegu
  - Daejeon
  - Goyang-si
  - Gyeonggi-do
  - Seoul

REFERENCES:
- See also: A comparative study of patient satisfaction between continued administration of previous antipsychotics versus switched administration to paliperidone ER in non-satisfied patients with previous antipsychotic drug — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=3450&filename=CR100782_CSR.pdf